CLINICAL TRIAL: NCT01931072
Title: The Effect of Exercise on Maximal Aerobic Capacity, DNA-methylation and Gene Expression in Healthy Elderly Men
Brief Title: Exercise-induced Changes in DNA-methylation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inconclusive results, large inter-individual variation, insufficient statistical power
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EPI-GEN100
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Healthy
Keywords: Exercise; High-intensity interval training; Moderate training; Healthy elderly; Skeletal muscle; DNA-methylation; Gene expression; subjects
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity interval training (Experimental): The High-intensity interval training group was instructed to complete exercise sessions of 4x4-minutes intervals at 85-95% of maximal heart rate, 3 times a week for 8 weeks. This type of exercise include 10 minutes warm-up, followed by four intervals of four minutes high-intensity (85-95% of HRmax), with three minutes active breaks (70% of HRmax) between each interval, and ending with seven minutes cool-down. An exercise session last for 42 minutes, where the participants should breathe heavily and feel exhausted four times.
  Interventions: Behavioral: High-intensity interval training
- Moderate training (Active Comparator): The moderate training group was instructed to complete exercise sessions of 50 minutes at 70% of maximal heart rate, 3 times a week for 8 weeks.
  Interventions: Behavioral: Moderate training
- Control (No Intervention): The control group followed the baseline and follow-up tests, and was asked to live normally and not change their dietary pattern or exercise habits during their participation in this project. Based on the well-known beneficial effects of exercise on general health, it was regarded unethical to demand the control group to desist from any types of physical activity during the project period. They got no further follow-up on exercise.

INTERVENTIONS:
Behavioral: High-intensity interval training — Interval training 3 times a week for 8 weeks
  Arms: High-intensity interval training
Behavioral: Moderate training — Moderate training 3 times a week for 8 weeks
  Arms: Moderate training

SUMMARY:
The purpose of the study was to investigate whether regular moderate- or high-intensity interval training can change the DNA methylation in a long-lasting state, and whether these changes affect the gene expression. In addition, the investigators will determine whether the intensity of the training could be an affecting factor of the possible DNA-methylation change as well. The null hypothesis was that no such exercise-induced changes occur.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 70-75 years old
* Signed written informed consent

Exclusion Criteria:

* Incompatible with exercise
* Known cardiac disease
* Active cancer
* Significant pulmonary disease
* Uncontrolled hypertension
* Use of blood thinning medicine (except Albyl-E)
* Drug abuse
* Alcohol abuse
* Finishing less than 80% of the exercise sessions (this complies to the training groups)

Ages: 70 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
DNA-methylation | 8 weeks
  From the skeletal muscle biopsies RNA and DNA was isolated, DNA was further bi-sulfite converted and DNA-methylation was analyzed using the Illumina HumanMethylation450 BeadChip. The RNA was further used for gene expression analyses by real-time RTqPCR.
Gene Expression | 8 weeks

SECONDARY OUTCOMES:
Maximal Aerobic Capacity | 8 weeks
  measured on treadmill at baseline and after eight weeks, also biopsies from Vastus lateralis were sampled.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisløff, Professor, Study Director — National Taiwan Normal University
Locations (1):
- Institute for Circulation and Medical Imaging, NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No